CLINICAL TRIAL: NCT03255603
Title: Gastrointestinal Assessment of Three Novel Resistant Starch Type IV
Brief Title: Gastrointestinal Assessment of Three Novel RS4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00069884
Record Dates: First submitted 2017-08-15; First posted 2017-08-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-05

CONDITIONS: Diet Modification
Keywords: Resistant Starch; Dietary Fiber; Gastrointestinal Microbiome; Gastrointestinal Tolerance
MeSH Terms: interventions — octenyl succinic anhydride-modified starch; Starch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Modified potato starch (Experimental): Modified potato starch is a resistant starch type IV and will be used as an experimental arm.
  Interventions: Other: Resistant Starch Type 4 Supplementation
- Modified corn starch (Experimental): Modified corn starch is a resistant starch type IV and will be used as an experimental arm.
  Interventions: Other: Resistant Starch Type 4 Supplementation
- Modified tapioca starch (Experimental): Modified tapioca starch is a resistant starch type IV and will be used as an experimental arm.
  Interventions: Other: Resistant Starch Type 4 Supplementation
- Corn starch (Placebo Comparator): Corn starch is digestible and will therefore will be used as a placebo control for the study.
  Interventions: Other: Digestible Starch Supplementation

INTERVENTIONS:
Other: Resistant Starch Type 4 Supplementation — Ten participants will supplement their normal dietary intake with RS4 daily for four consecutive weeks, with each week the amount of RS4 provided being increased (10 g, 20 g, 35 g and 50 g/day).
  Other Names: Modified potato starch
  Arms: Modified potato starch
Other: Resistant Starch Type 4 Supplementation — Ten participants will supplement their normal dietary intake with RS4 daily for four consecutive weeks, with each week the amount of RS4 provided being increased (10 g, 20 g, 35 g and 50 g/day).
  Other Names: Modified corn starch
  Arms: Modified corn starch
Other: Resistant Starch Type 4 Supplementation — Ten participants will supplement their normal dietary intake with RS4 daily for four consecutive weeks, with each week the amount of RS4 provided being increased (10 g, 20 g, 35 g and 50 g/day).
  Other Names: Modified tapioca starch
  Arms: Modified tapioca starch
Other: Digestible Starch Supplementation — Ten participants will supplement their normal dietary intake with digestible starch daily for four consecutive weeks, with each week the amount of starch provided being increased.
  Other Names: Corn starch
  Arms: Corn starch

SUMMARY:
The rates of chronic diseases like obesity, diabetes, and heart disease are rising across the world. This is especially true in industrialized countries like Canada and the USA. Even though there are many possible causes for these increases. One prominent cause is our refined diet, which greatly lacks dietary fiber. This 'fiber gap' between the amount of fiber actually eaten and the amount that should be eaten is likely promoting these diseases.

It is known that a high fiber diet can benefit health and the health of the gut bacteria. It is also know that these gut microbes can help cause and prevent diseases. When fiber is eaten, it gets broken down not by us, but by our gut microbes. During this process by-products called short-chain fatty acids (SCFA) are made. These SCFA have been shown to promote health. Therefore, it is thought that fiber changes the gut microbes to produce more SCFA, which may improve overall health.

In order to aid our microbes and improve our health we need to find ways to reduce this 'fiber gap'. One possibility is to add fiber to our refined diet. To do so we must first learn how different fibers perform in our gut. This includes how our gut tolerates increasing amounts of fiber, and how our microbes respond. The purpose of this study is to learn how different types of resistant starch perform in our gut, including gastrointestinal tolerance. By doing so we will determine the ideal dose and type of these fibers to use in future studies.

DETAILED DESCRIPTION:
The investigators propose a 4 week gastrointestinal (GI) assessment study to determine both the ideal dose and type of resistant starch to use in future studies. The following specific aims are offered:

AIM 1: GI Tolerance. Preform a randomized, placebo-controlled, double-blind, parallel-four-arm human intervention study to assess the GI tolerance of 3 novel resistant starch type IV (RS4) at dose up to 50 g per day.

Interested participants will be asked to attend a screening visit at Human Nutrition Research Unit, where lifestyle and anthropometric information will be collected to determine eligibility. Eligible participants (N = 40) will be stratified based on gender and randomly assigned to 1 of 4 groups, where they will be asked to supplement their diet for 4 weeks with either a RS4 (experimental arms) or a digestible starch (control arm). The weight of total starch (digestible plus RS) provided in each experimental arm will be dependent on the purity of the individual RS4 products. Subjects will supplement their diet with 10 g, 20 g, 35 g and 50 g of total dietary fiber (as RS) daily over the course of weeks 1, 2, 3 and 4, respectively. The amount of digestible starch provided in the control arm will be equal to the mean amount of total starch provided across the 3 experimental arms. All starch products will be provided in powder form.

Methodologies previously described by Maki et al. will be employed to evaluate the overall GI tolerance of the RS4 products by assessing changes in GI symptom, bowel movement frequency, and bowel movement consistency, and by comparing these changes to those changes observed in the control arm (digestible starch - Maki et al., Int J Food Sci Nutr, 2013). Participants will keep a daily study journal, which included a bowel habits questionnaire, over the course of the 4 week study, and they will also complete weekly GI tolerance and satiety questionnaires during their weekly study visits. Participants will also be asked to complete two 24-h recalls, both prior to starting the dietary intervention and during week 4. All 24-h recalls will be completed online through the Canadian Automated Self-Administered 24h (ASA24) recall system.

AIM 2: Evaluate prebiotic and dose dependent effect on the microbiome. Evaluate the effect of the 3 distinct RS4 types on gut microbiota composition and structure in a dose dependent manner.

Fecal samples will be collected at baseline and at the end of each intervention week (weeks 1-4). Fecal samples will be used to both characterize the fecal microbial community via 16S ribosomal RNA next-generation sequencing, and to quantify fecal short-chain fatty acid concentrations via gas chromatography. Short-term characterization of the fecal microbiome will provide a systematic assessment of the individualized response between 3 structurally distinct types of RS4, while further allowing an intricate assessment of the prebiotic dose effect upon significantly increasing the dose of RS towards 50 g per day. This analysis will provide critical information on how distinct types of RS4 shape the gut microbiome in humans, and which dose is necessary to achieve such effects.

ELIGIBILITY:
Inclusion Criteria:

* men and pre-menopausal, non-pregnant or non-lactating women
* non-vegetarian
* non-smoking
* alcohol intake ≤8 drinks/week
* ≤5 h/week of moderate-vigorous exercise

Exclusion Criteria:

* acute or chronic GI illnesses, conditions, or issues
* history of GI surgical intervention
* chronic or current use of anti-hypertensive, lipid-lowering, anti-diabetic, analgesic, or laxative medications
* antibiotic treatment in the last 3 months
* use of fiber or probiotics supplements
* allergies or intolerances to fiber sources

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-12-22 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Tolerance | 4-week period
  Gastrointestinal tolerance will be assessed at weeks 0-4 of fiber intervention with a weekly gastrointestinal tolerability questionnaire.

SECONDARY OUTCOMES:
Gastrointestinal Habits | 4-week period
  Gastrointestinal habits will be assessed at weeks 0-4 of fiber intervention with a weekly bowel habit questionnaire.
Gastrointestinal Microbiome Composition | 4-week period
  Fecal microbial composition will be characterized at weeks 0-4 of fiber intervention by 16S rRNA sequencing.
Gastrointestinal Microbiome Function | 4-week period
  Fecal microbial function will be assessed at weeks 0-4 of fiber intervention through fecal SCFA concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Walter, PhD, Principal Investigator — University of Alberta
Locations (1):
- Alberta Diabetes Institute Clinical Research Unit, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No